CLINICAL TRIAL: NCT03038087
Title: An Early Feasibility Study to Evaluate the User Interfaces and Sensitivity of the SENSE Device in Patients With Intracranial Hemorrhage
Brief Title: A Study to Test the SENSE Device in Patients With Intracranial Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sense Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SENSE-001
Record Dates: First submitted 2017-01-19; First posted 2017-01-31 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Intracerebral Hemorrhage; Stroke, Acute; Stroke Hemorrhagic
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SENSE Device Monitoring in ICH Patients (Experimental): The SENSE device transmits a low power tailored electro-magnetic (EM) pulse in the radio-frequency range across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage. The device consists of two parts:
  1. A molded plastic headpiece containing the antenna array, and
  2. A processing control unit that contains:
     1. The driving electronics for the array;
     2. A spectrum analyzer coupled with a computer; and,
     3. The operating software that controls the device function and data acquisition, processing and archiving.
  For this study, the research personnel will place the headset over the subject's head. The headset will be sized to fit snuggly. Each headset is marked with a unique headset identification number. The patient-contacting components of the molded plastic form are made from a medical grade (USP Class VI), biocompatible plastic and foam.
  Interventions: Device: SENSE Device

INTERVENTIONS:
Device: SENSE Device — The SENSE device transmits a low power tailored electro-magnetic pulse across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage. The device consists of two parts:
  1. A molded plastic headpiece containing the antenna array, and
  2. A processing control unit.
  The SENSE device will be placed on the subject within 15 minutes of a baseline head CT, or as soon as practicable. The SENSE device will be set to scan every 10 minutes until the device is removed after completion of the SENSE measurement corresponding to the 72 hour CT scan. The investigator will be blinded to the data collected from the SENSE device.

SUMMARY:
The purpose of this research study is to find out whether a device for monitoring bleeding in patients with acute hemorrhagic stroke will show similar findings as CT scans performed to evaluate the stroke.

DETAILED DESCRIPTION:
This will be a prospective, observational, single site, first-in-man study of the SENSE device in up to 10 study subjects with primary spontaneous ICH. The treating clinicians will be blinded to the data collection and SENSE device scanning as described below.

All eligible subjects must have the diagnostic head CT scan (CT) demonstrating hemorrhage performed within 6 hours of symptom onset. While ICH and TBI patients may be evaluated in future studies, this early feasibility study is limited to primary spontaneous ICH patients only, given the relative homogeneity of this population compared with the TBI population.

Eligible subjects or legally authorized representatives will be approached for enrollment. After obtaining informed consent to participate in the study, a baseline study head CT will be performed to establish the hemorrhage volume; and the SENSE device will be placed on the subject within 15 minutes of this CT, or as soon as practicable, for initiation of monitoring. This repeat CT (after the diagnostic CT) is necessary since hemorrhage expansion (HE) occurs early in the clinical course, and the hemorrhage volume may have changed between the diagnostic CT and placement of the SENSE monitor.

After enrollment, routine clinical management will ensue in the emergency department (ED), hospital ward or intensive care unit (ICU) as appropriate. A standard of care head CT to evaluate for HE will be performed at 12 (±6) hours after the baseline study head CT. Finally, a study head CT will be performed at 72 (±12) hours to evaluate cerebral edema. Any head CT performed for clinical deterioration as standard of care between the baseline and 72 hour study CTs will also be collected and analyzed.

The SENSE device will be placed on the subject's head, and two small ink dots will be marked on the head corresponding to a known location on the device to allow for the device to be removed and replaced consistently throughout testing. The SENSE device will be set to scan every 10 minutes until the device is removed after completion of the SENSE measurement corresponding to the 72 hour CT scan. If the SENSE device is removed to perform the CT or SENSE monitoring is temporarily suspended, the SENSE device will be replaced; and SENSE monitoring will resume within 15 minutes, or as soon as practicable, after each CT scan. A SENSE measurement obtained within 15 minutes of each CT scan, or as soon as practicable thereafter, will be used for comparison with data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 22 years and older
2. Diagnostic head CT scan within 24 hours of primary spontaneous ICH symptom onset
3. ICH >3mL and <90mL, as measured by the ABC method
4. Signed written informed consent by study subject or, if subject is unable, by subject's next of kin or legal guardian
5. Willingness and ability to comply with schedule for study procedures

Exclusion Criteria:

1. Female patients who are pregnant or lactating
2. Patients with any history of seizure or seizure at stroke onset
3. Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for the SENSE device monitoring or study participation or may confound the outcome of the study
4. Any intraventricular hemorrhage on the diagnostic (pre-enrollment) CT with planned placement of an intraventricular catheter
5. Secondary cause of ICH suspected (e.g., arteriovenous malformation, cavernoma, aneurysm, hemorrhagic transformation ischemic stroke, venous sinus thrombosis, trauma)
6. Planned withdrawal of care within 24 hours of enrollment
7. Planned surgical evacuation within 24 hours of enrollment
8. Current participation in a medical or surgical interventional clinical trial
9. Presence of subdural, epidural or aneurysmal subarachnoid hemorrhage on diagnostic scan
10. Planned continued use or prescribed use during the study of medications that, in the investigator's best clinical judgment, are known or suspected to lower the seizure threshold
11. Planned continued use of medications that, in the investigator's best clinical judgment, could increase the chances for subsequent uncontrolled hemorrhage
12. Planned or current use of continuous EEG monitoring

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Knight, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SENSE Device Monitoring in ICH Patients: The SENSE device transmits a low power tailored electro-magnetic (EM) pulse in the radio-frequency range across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage. The device consists of two parts:
  1. A molded plastic headpiece containing the antenna array, and
  2. A processing control unit that contains:
     1. The driving electronics for the array;
     2. A spectrum analyzer coupled with a computer; and,
     3. The operating software that controls the device function and data acquisition, processing and archiving.
  For this study, the research personnel will place the headset over the subject's head. The headset will be sized to fit snuggly. Each headset is marked with a unique headset identification number. The patient-contacting components of the molded plastic form are made from a medical grade (USP Class VI), biocompatible plastic and foam.
  The SENSE device will be placed on the subject within 15 minutes of a baseline head CT, or as soon as practicable. The SENSE device will be set to scan every 10 minutes until the device is removed after completion of the SENSE measurement corresponding to the 72 hour CT scan. The investigator will be blinded to the data collected from the SENSE device.
Period: Overall Study
Arm/Group | SENSE Device Monitoring in ICH Patients
Started | 10
Completed | 9
Not Completed | 1
Not completed — lost data | 1

BASELINE CHARACTERISTICS:
Arm/Group | SENSE Device Monitoring in ICH Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 57 [43 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Serious Device-related Adverse Events
Description: Number of subjects who experienced a serious device-related adverse event or seizure.
Time Frame: Up to 6 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Who Experienced Serious Device-related Adverse Events or Seizure.: The number of subjects who experienced a device related serious AE and/or seizures will be tabulated and summarized.
Arm/Group | Subjects Who Experienced Serious Device-related Adverse Events or Seizure.
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Number of Patients Correctly Identified by SENSE With Hemorrhage Expansion (HE) or no Hemorrhage Expansion (NHE) Within 12 Hours.
Description: The SENSE device continuously monitored patients for hemorrhage expansion (HE) defined as a greater than 3 ml increase in ICH volume. ICH volumes were determined from the CT scans by a neuroradiologist. The concordance of SENSE determination of HE or NHE with the CT results was determined.
Time Frame: 12 Hours
Population: Study subjects were drawn from patients suffering from ICH. These patients either presented or transferred to a large, urban, comprehensive stroke center.
Measure: Count of Participants; unit: Participants
Groups:
- ICH Patients With Hemorrhage Expansion: The primary aim was to determine determine the ability of the SENSE device to detect a clinically significant (>= 3 ml) hemorrhage expansion in ICH patients. ICH volume was determined by CT measurements at 0, 12, and up to 72 hours (if available).
Arm/Group | ICH Patients With Hemorrhage Expansion
Number analyzed (Participants) | 9
Participants
  ICH Subjects with expansion: number analyzed (Participants) | 2
  ICH Subjects with expansion | 2
  ICH Patients without expansion: number analyzed (Participants) | 7
  ICH Patients without expansion | 7

3. Secondary Outcome: Feasibility of the SENSE Device in a Clinical Environment
Description: Number of patients where data was successfully acquired, downloaded, and analyzed.
Time Frame: Up to 72 Hours
Population: Patients were monitored with SENSE for an average of 60 (range: 23-72) hours. There were no serious adverse events. Minor adverse events were predominantly minor skin and nose irritation from the nosepiece of the headset. 1 Patient did not finish the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SENSE Device Monitoring in ICH Patients
Number analyzed (Participants) | 10
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SENSE Device Monitoring in ICH Patients
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SENSE Device Monitoring in ICH Patients (N=10)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Redness caused by device pressing on skin and bridge of nose
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT03038087/Prot_SAP_001.pdf